CLINICAL TRIAL: NCT06193603
Title: Effectiveness of Cupping Therapy in Patients With Chronic Nonspecific Low Back Pain: a Randomized Sham-controlled Trial
Brief Title: Cupping Therapy in Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.IUMS.REC.1401.455
Record Dates: First submitted 2023-12-09; First posted 2024-01-05 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low-back Pain; Chronic Non-specific Low Back Pain; Low Back Pain; Cupping Therapy
Keywords: Chronic non-specific low back pain; Cupping therapy; Randomized sham-controlled trial
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant) Participants in the control group will undergo a similar procedure to those in the intervention group. Two cups will be placed on the lumbar region, but the sham cups will have small holes (<2mm in diameter) to release negative pressure quickly. Additionally, to reduce bias, the data analyst will be blinded to the group assignments of the participants. Each participant will be identified by a unique numerical code to maintain anonymity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- True dry cupping therapy (Experimental): Participants in the true dry cupping therapy group, who have chronic non-specific low back pain, will receive a combination of dry cupping therapy and routine physiotherapy. During the dry cupping therapy sessions, two cups will be applied to the lumbar region and moved in an up-down and down-up direction.
  Interventions: Other: True dry cupping therapy
- Sham cupping therapy (Sham Comparator): Participants in the sham cupping therapy group, who have chronic non-specific low back pain, will undergo a combination of sham cupping therapy and routine physiotherapy. During the sham cupping therapy sessions, two cups with small holes will be placed stationary on the lumbar region.
  Interventions: Other: Sham cupping therapy

INTERVENTIONS:
Other: True dry cupping therapy — In the intervention group, participants will lie in a prone position, and the lumbar area between L1-L5 will be oiled. Two cups with a diameter of 4.5-5 cm will be placed bilaterally, parallel to the lumbar spine. The therapist will perform 5 minutes of dry cupping therapy, moving the cups up and down using both hands. Participants will also receive routine physiotherapy, including a 20-minute session of transcutaneous electrical stimulation with a frequency of 100 pulses per second and a duration of 60 microseconds. The stimulation intensity will be adjusted for sensory stimulus. Stabilization exercises like abdominal hollowing and bridging will be included. The treatment will consist of 10 sessions, three times per week.
  Arms: True dry cupping therapy
Other: Sham cupping therapy — In the control group, participants will lie in a prone position, and the lumbar area between L1-L5 will be oiled. Two cups with a diameter of 4.5-5 cm will be placed bilaterally, parallel to the lumbar spine. However, unlike the intervention group, the cups in the control group will not be moved and will remain stationary for 5 minutes. The cups will have small holes (<2mm in diameter) to release negative pressure quickly. Double-sided tapes will be used to secure the cups and maintain contact with the skin.
  Arms: Sham cupping therapy

SUMMARY:
Chronic non-specific low back pain is a common condition that can cause disability, physical and psychological impairment, limitations in daily activities, and participation restrictions. It also has significant economic and social impacts. Clinical guidelines recommend non-pharmacological interventions as the first-line treatment, including exercises, psychological therapies, and multidisciplinary rehabilitation. Pharmacological therapies are used when non-pharmacological approaches are not effective. Alternative therapies like cupping therapy have gained attention, but their efficacy is still debated due to limited high-quality studies. Further research is needed to determine the true benefits and effectiveness of cupping therapy in managing chronic low back pain. A recent study found that dry cupping therapy was not superior to sham cupping in improving pain, physical function, mobility, quality of life, psychological symptoms, or medication use in individuals with chronic non-specific low back pain. However, it's important to note that the study used dry cupping therapy in isolation, which may not reflect typical clinical practice. Well-designed clinical trials can provide a better understanding of the potential impact of cupping therapy on various aspects of chronic low back pain. Hence, the primary goal of this randomized clinical trial is to compare the effectiveness of true cupping therapy combined with routine physiotherapy versus sham cupping therapy combined with routine physiotherapy in patients suffering from chronic non-specific low back pain. The study aims to address the following key questions:

* Does true dry cupping therapy, when combined with routine physiotherapy, provide greater improvement in pain and functional disability for patients with chronic non-specific low back pain?
* Does true dry cupping therapy, when combined with routine physiotherapy, result in a higher improvement in quality of life for patients with chronic non-specific low back pain?

Participants in the intervention group will undergo 10 sessions of dry cupping therapy, with each session lasting 5 minutes and conducted three times per week. During the sessions, the therapist will move the cups longitudinally in upward-downward and downward-upward directions. In the control group, participants will assume the same positions as the intervention group, but two cups with small holes (<2mm in diameter) will be used to release negative pressure within seconds.

DETAILED DESCRIPTION:
RESEARCH OBJECTIVE:

The primary objective of this study is to examine the efficacy of true dry cupping therapy, in combination with routine physiotherapy, in comparison to sham dry cupping therapy, in combination with routine physiotherapy, for managing pain intensity and functional disability in individuals with chronic non-specific low back pain. The secondary objective is to evaluate the impact of 10 treatment sessions on the quality of life of patients with chronic non-specific low back pain.

RESEARCH DESIGN:

This study is a randomized, single-blind, sham-controlled trial conducted at two centers. The allocation ratio is 1:1, with a total of 80 participants with hypertrophic scar tissue. Random assignment to two groups of equal size will be done using the permuted block randomization method, utilizing four-letter blocks (A and B). The random treatment list will be placed in sealed and numbered envelopes, with letter A representing true dry cupping therapy and letter B representing sham dry cupping therapy. The random assignment process will be conducted by an individual outside the research team prior to the commencement of the study.

PROCEDURE:

At the beginning of the study, potential participants will undergo an assessment to determine their eligibility based on specific criteria. Once confirmed by an orthopedic surgeon, participants will be enrolled in the study. Eligible participants will be asked to complete an intake form, providing demographic data such as age, gender, height, weight, occupation, and information regarding major confounding variables like smoking and depression that may affect low back pain. Following that, participants will be requested to complete questionnaires assessing pain intensity, functional disability, and quality of life.

INTERVENTION:

After the baseline assessment, the principal investigator will administer dry cupping therapy to the intervention group consisting of 24 enrolled patients. The participants in this group will be asked to lie in a prone position, and the lumbar area between L1-L5 will be oiled. Two cups with a diameter of 4.5-5 cm will be placed bilaterally parallel to the lumbar spine vertebrae. The therapist will then perform dry cupping therapy by applying two suctions and moving the cups in an up-down and down-up direction for 5 minutes using both hands.

In contrast, the control group will assume the same positions as the intervention group, but the cups will be placed stationary for 5 minutes only. The cups in the control group will have small holes with a diameter of less than 2mm to release negative pressure within seconds. Double-sided tapes will be used to secure the cups and maintain contact with the skin.

Both groups will undergo routine physiotherapy, which includes a 20-minute session of transcutaneous electrical stimulation. The stimulation will be set at a frequency of 100 pulses per second and a duration of 60 microseconds. The intensity of the stimulation will be gradually adjusted until participants experience a sensory stimulus during the 20-minute session. Stabilization exercises such as abdominal hollowing and bridging exercises will also be included in the treatment.

The entire treatment duration will consist of 10 sessions, conducted three times per week.

REASSESSMENT:

After the interventions, measures of the primary and secondary outcomes will be collected immediately and two weeks after the final treatment session to evaluate the effectiveness of the cupping therapy intervention. Additionally, any adverse events following the cupping therapy procedures and adherence to the treatment will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific low back pain lasting for a minimum of 3 months.
* The pain intensity is rated between 3 and 6 on the visual analog scale.
* The body mass index falls between 19 and 23.
* No restrictions for therapeutic exercise and electrotherapy.

Exclusion Criteria:

* The presence of comorbidities such as diabetes and cardiovascular problems.
* The presence of spinal column deviations, such as scoliosis, is observed.
* Signs of serious pathology of the spine (eg, fractures, inflammatory diseases, infection or tumours).
* Consecutive absence of more than three sessions.
* Patients' dissatisfaction with their participation in the study
* Individuals who have been treated with cupping in the past.
* Neurological, vestibular, visual or auditory deficits.
* Currently performing physical therapy.
* Irradiated lumbar or sacroiliac pain.
* Fibromyalgia

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline at 4-week and 6-week
  The Numeric Pain Rating Scale (NPRS) will be utilized to assess changes in pain levels. This scale ranges from 0 to 100, with 0 representing no pain and 100 representing the maximum level of pain experienced by the patient. The NPRS has demonstrated responsiveness in measuring pain levels among individuals with low back pain.
Functional disability | Change from baseline at 4-week and 6-week
  The Persian version of the Oswestry Disability Index (ODI) will be employed to assess changes in functional disability. This questionnaire comprises 10 activities of daily living and yields a total score ranging from 0 to 100. A score below 25 indicates minimal disability, while scores between 25 and 50 represent moderate disability. Scores between 50 and 75 indicate severe disability, and scores between 75 and 100 reflect acute disability. The Persian version of this questionnaire has been previously validated and shown to be reliable in previous studies.

SECONDARY OUTCOMES:
Quality of life assessment | Change from baseline at 4-week and 6-week
  The self-reported quality of life based on the 36-Item Short-Form Health Survey (SF-36) will be assessed. This questionnaire consists of 36 items divided into 8 subscales: Physical Functioning, Role limitations due to physical problems, Bodily Pain, Vitality, General Health, Social Functioning, Role limitations due to emotional problems, and Mental Health. The scale ranges from 0 to 100. 0 denotes minimal quality of life and 100 denotes maximum quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammadreza Pourahmadi, Principal Investigator — Iran University of Medical Sciences
Locations (1):
- Iran University of Medical Sciences, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Almeida Silva HJ, Barbosa GM, Scattone Silva R, Saragiotto BT, Oliveira JMP, Pinheiro YT, Lins CAA, de Souza MC. Dry cupping therapy is not superior to sham cupping to improve clinical outcomes in people with non-specific chronic low back pain: a randomised trial. J Physiother. 2021 Apr;67(2):132-139. doi: 10.1016/j.jphys.2021.02.013. Epub 2021 Mar 20. PMID 33757719
- [Background] Silva HJA, Saragiotto BT, Silva RS, Lins CAA, de Souza MC. Dry cupping in the treatment of individuals with non-specific chronic low back pain: a protocol for a placebo-controlled, randomised, double-blind study. BMJ Open. 2019 Dec 22;9(12):e032416. doi: 10.1136/bmjopen-2019-032416. PMID 31871257
- [Background] Moura CC, Chaves ECL, Cardoso ACLR, Nogueira DA, Correa HP, Chianca TCM. Cupping therapy and chronic back pain: systematic review and meta-analysis. Rev Lat Am Enfermagem. 2018 Nov 14;26:e3094. doi: 10.1590/1518-8345.2888.3094. PMID 30462793
- [Background] Huang CY, Choong MY, Li TS. Effectiveness of cupping therapy for low back pain: a systematic review. Acupunct Med. 2013 Sep;31(3):336-7. doi: 10.1136/acupmed-2013-010385. Epub 2013 Jul 25. No abstract available. PMID 23886511
- [Background] Wang L, Cai Z, Li X, Zhu A. Efficacy of cupping therapy on pain outcomes: an evidence-mapping study. Front Neurol. 2023 Oct 26;14:1266712. doi: 10.3389/fneur.2023.1266712. eCollection 2023. PMID 37965178
- [Background] Volpato MP, Breda ICA, de Carvalho RC, de Castro Moura C, Ferreira LL, Silva ML, Silva JRT. Single Cupping Thearpy Session Improves Pain, Sleep, and Disability in Patients with Nonspecific Chronic Low Back Pain. J Acupunct Meridian Stud. 2020 Apr;13(2):48-52. doi: 10.1016/j.jams.2019.11.004. Epub 2019 Nov 21. PMID 31760207
- [Background] Teut M, Ullmann A, Ortiz M, Rotter G, Binting S, Cree M, Lotz F, Roll S, Brinkhaus B. Pulsatile dry cupping in chronic low back pain - a randomized three-armed controlled clinical trial. BMC Complement Altern Med. 2018 Apr 2;18(1):115. doi: 10.1186/s12906-018-2187-8. PMID 29609566
- [Background] Salemi MM, Gomes VMDSA, Bezerra LMR, Melo TMS, Alencar GG, Montenegro IHPM, Calado APM, Montenegro EJN, Siqueira GR. Effect of Dry Cupping Therapy on Pain and Functional Disability in Persistent Non-Specific Low Back Pain: A Randomized Controlled Clinical Trial. J Acupunct Meridian Stud. 2021 Dec 31;14(6):219-230. doi: 10.51507/j.jams.2021.14.6.219. PMID 35770601
- See also: Related Info — http://dergipark.org.tr/en/pub/omujecm/issue/73188/1121925